CLINICAL TRIAL: NCT06635434
Title: Feasibility of a Dual English/Spanish Mobile Augmented Reality Pain Assessment App to Reduce Postoperative Prescription Opioid Use in Hispanic/Latino Pediatric and Adolescent Cancer Patients
Brief Title: An English/Spanish Mobile Augmented Reality Pain Assessment App for Hispanic/Latino Pediatric Cancer Patients
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: ALTality, Inc. (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1R43DA057744-01 (NIH)
Record Dates: First submitted 2024-09-19; First posted 2024-10-10 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Pain; Pediatric Cancer
MeSH Terms: conditions — Pain; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Augmented reality-enabled pain assessment deployed on a mobile (Experimental): Age-stratified (age 7-11 and age 12-17 years old) augmented reality app to evaluate for pain and opioid-related adverse events with equivalent English and Spanish text, audio, and narration
  Interventions: Device: AR Pain assessment

INTERVENTIONS:
Device: AR Pain assessment — Age-stratified (age 7-11 and age 12-17 years old) augmented reality app to evaluate for pain and opioid-related adverse events with equivalent English and Spanish text, audio, and narration

SUMMARY:
In this SBIR, ALTality, Inc. ("SpellBound") will assess the feasibility of a dual English/Spanish language augmented reality(AR)-enabled tool for assessing inpatient postoperative pain/nausea/vomiting in Hispanic/Latino children and adolescents with cancer in collaboration with bilingual Spanish-speaking anesthesiologists at the MD Anderson Cancer Center. If successful, the AR app will be an immediately implementable and commercially viable method of providing Hispanic/Latino pediatric cancer patients with limited English proficiency an adjunctive tool to overcome infrastructural barriers to receiving translation services in acute care settings that put them at higher risk of under and/or overtreatment of pain by prescription opioids and future prescription opioid dependency and misuse, at no cost to them or their families.

ELIGIBILITY:
Inclusion Criteria:

* ages 7-17 years old
* child able to provide assent, and a legal guardian able to provide informed consent
* current diagnosis of pediatric cancer
* undergoing surgery for cancer treatment requiring postoperative inpatient hospitalization
* prescribed or expected to be prescribed opioids during inpatient perioperative period
* sufficient mental capacity to comprehend and interact with the game in English or Spanish.

Exclusion Criteria:

* the inability to play with the SpellBound app from English or Spanish instructions
* daily opioid use within 30 days prior to surgery
* any concerns from the treatment team.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2023-02-05 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Primary; Percent of enrolled patients who activated/used the app during the PACU stay | immediately after the intervention/procedure/surgery
  Feasibility measured as activation/usage of the app recorded by the device ID for each patient

SECONDARY OUTCOMES:
Total time spent playing on the AR app during the PACU stay | immediately after the intervention/procedure/surgery
  Length of time (minutes) of app usage recorded by the device ID for each patient
Recorded responses about pain assessment from the app | immediately after the intervention/procedure/surgery
  Pain scale score in English or Spanish through the app
Recorded responses about nausea/vomit assessment from the app | immediately after the intervention/procedure/surgery
  Baxter animated retching scale score in English or Spanish through the app
Inpatient opioid consumption | immediately after the intervention/procedure/surgery
  Calculated as morphine equivalent dose of all opioids given
Length of stay | immediately after the intervention/procedure/surgery
  Total time (minutes) spent in the PACU after surgery
Quality of life survey | immediately after the intervention/procedure/surgery
  PedsQL survey administered to child and/or adult caregiver stratified by age
Rate of opioid prescription | immediately after the intervention/procedure/surgery
  The percentage of patients with opioid prescriptions at the time of discharge from the electronic health record
Patient/caregiver satisfaction survey | immediately after the intervention/procedure/surgery
  Asked to the patient/caregiver by the study team - 1) How satisfied were you with regards to your pain management in PACU?, 2) How satisfied were you with regards to your nausea management in PACU?, 3) How satisfied were you with the use of the AR app to help assess your pain and nausea?

CONTACTS AND LOCATIONS:
Overall Officials: Christina York, Principal Investigator — ALTality, Inc.
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Pediatric cancer diagnoses are rare and by definition could identify individual patients and violate patient privacy.

REFERENCES:
- [Background] Kamaladevi RK, Elakkumanan LB, Regmi S. Smart Anesthesia-Another Way of Communication During Emergence from Anesthesia Using a Smartphone. Anesth Analg. 2016 Aug;123(2):518. doi: 10.1213/ANE.0000000000001400. No abstract available. PMID 27258079
- [Background] Gaither JR, Leventhal JM, Ryan SA, Camenga DR. National Trends in Hospitalizations for Opioid Poisonings Among Children and Adolescents, 1997 to 2012. JAMA Pediatr. 2016 Dec 1;170(12):1195-1201. doi: 10.1001/jamapediatrics.2016.2154. PMID 27802492